CLINICAL TRIAL: NCT04129489
Title: A Phase 2a Open Label, Single Arm Study to Evaluate the Safety and Efficacy of Cannabidiol Only as Maintenance Therapy and Steroid Sparing in Patients With Stable Autoimmune Hepatitis
Brief Title: A Phase 2a Study to Evaluate the Safety and Efficacy of Cannabidiol Only as Maintenance Therapy and Steroid Sparing in Patients With Stable Autoimmune Hepatitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low recruitment
Sponsor: Stero Biotechs Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ST-AH-01
Record Dates: First submitted 2019-03-18; First posted 2019-10-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Autoimmune Hepatitis
MeSH Terms: conditions — Hepatitis, Autoimmune | interventions — Cannabidiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sintetic Cannabidiol (Experimental): Synthetic Cannabidiol, dissolved in pharmaceutical grade olive oil at a concentration of 5% will be administered orally twice a day
  Interventions: Drug: Cannabidiol

INTERVENTIONS:
Drug: Cannabidiol — Synthetic Cannabidiol, dissolved in pharmaceutical grade olive oil at a concentration of 5% will be administered orally

SUMMARY:
Subjects with stable autoimmune hepatitis disease currently being administered corticosteroids with or without azathioprine (AZA) treatment will be be treated with Cannabidiol instead of standard of care treatment with corticosteroids

DETAILED DESCRIPTION:
Patients will be included if they are in stable remission with a prednisone at the lower stable dose to maintain remission with or without azathioprine , Budesonide with or without azathioprine or azathioprine alone for at least 24 months.

Patient will be switch from standard of care to treatment with Cannabidiol for 12 months. They will receive increasing doses of Cannabidiol over a period of one month. Dosage will start at 25 mg Cannabidiol twice a day and will be increased every seven days, if no side effects are observed, to 50 mg, 100 mg and finally to 150 mg Cannabidiol twice a day respectively, as detailed below.

At the end of this month, if the 150 mg twice a day dose level is deemed safe for one week, the standard of care will be stopped at once and patients will continue receiving only Cannabidiol 150 mg twice a day for an additional period of 11 months.

The patient will be offered to undergo liver biopsy in the screening period to prove histological remission along with the biochemical remission (not mandatory for inclusion).

After 12 months of treatment with Cannabidiol all patient will undergo liver biopsy for confirmation of histological remission and then the treatment will be stopped as for physician decision and guidelines of treatment of autoimmune hepatitis disease.

In any case of flare defined as elevation in liver enzymes and immunoglobulins in consecutive blood test the patient will reintroduced for standard of care treatment at a dosage as of investigator decision and the Cannabidiol will be discontinued.

The patient will be withdrawn from the study but will continue follow up until returning to stable inactive disease as define as normalization of liver enzymes and immunoglobulin level in consecutive blood tests.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed chronic hepatitis
2. Age ≥18 years
3. Subject able to provide written informed consent
4. Stable disease for 24 months
5. Currently being administered prednisone (with or without azathioprine) therapy at the lower stable dose to maintain remission or Budesonide (with or without azathioprine) therapy at the lower stable dose to maintain remission or azathioprine alone.
6. ALT ≤ 30 U/L in men and ≤19 U/L in women
7. IgG < 1450 mg/dL
8. Non-pregnant women (via negative pregnancy test) and women with no intention to become pregnant during the term of the trial or three months after cessation of CBD treatment

Exclusion Criteria:

1. Viral Hepatitis (HAV, HBV, HCV)
2. HIV
3. Serious psychiatric or psychological disorders
4. Active consumption of illicit drugs including cannabis or derivatives (at least 1 month before study start)
5. Overlap disease with Primary Biliary Cholangitis or Primary Sclerosing Cholangitis
6. IgG4 related Autoimmune Hepatitis
7. Transplant patients
8. Patients with significant cardiac, respiratory or active malignance disease comorbidities.
9. Renal comorbidity: eGFR < 30 mL/min/1.73 m2 (note: CKD Grade 4 is defined as eGFR 15-29 mL/min/1.73 m2)
10. Cirrhosis
11. Patients treated with corticoids for other indication except Autoimmune Hepatitis
12. Patient that are taking immunomodulatory medications for other indication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-02-07 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with biochemical and histological remission | 12 month
  biochemical and histological data will be collected during the study
Number of patients who experience Cannabidiol relates adverse events | 12 month
  Adverse events will be recorded during the study
Proportion of patients with flare up of hepatitis | 12 month
  record of disease flare will be collected during the study

CONTACTS AND LOCATIONS:
Locations (1):
- Belinson Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: Undecided